CLINICAL TRIAL: NCT02337998
Title: The Effect of Load Carriage on Upper Limb Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Gabriel Zeilig, Director, Department of Neurological Rehabilitation, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1593-14-SMC
Record Dates: First submitted 2015-01-06; First posted 2015-01-14 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Healthy
Keywords: Neurology; Sports Medicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy men (Experimental): each individual will serve as his own control by comparing baseline values to post intervention values
  Interventions: Other: load carriage

INTERVENTIONS:
Other: load carriage

SUMMARY:
Purpose: Quantify the relationship between brachial plexus deformations caused by backpack carriage and upper extremity performance.

Significance of expected results:

The study will allow to quantify the effect of load carriage on both neural and vascular function parameters.

Study plan The effect of nerve strain on neural function: based on the strains obtained for each load from computational simulation, and from animal studies published in the literature, the expected neural function, (e.g., motor and sensory) dysfunction will be estimated.

Following signing an informed consent form, 12 young adult subjects (18-35 years) will don a military backpack loaded with 25-40 kg. Each volunteer will undergo the following test at baseline, following 45 min exposure, and following 15 min of recovery:

1. Index finger microvascular flow will be measured by photoplethysmography (PPG).
2. Sensory measurement at the finger; Light touch threshold will be measured by mechanical stimulation that will be applied using Von Frey Filaments of the Semmes-Weinstein Monofilament (SWM) type.
3. Forearm thermal sensation threshold; As a measure of sensory function in the forearm, cold and warm sensation thresholds will be measured with a computerized quantitative thermal sensory device.

   Immediately following the 45 min loading exposure, the fine motor function of the index finger will be tested by the following procedures (in an unloaded condition):
4. Index finger motor function; Force application profile during a trigger press will be measured using a force sensor located on a trigger of a dummy weapon simulator. Force application rate, peak force, and press-to-press peak force variability will be measured based on 10 trigger presses.
5. Accuracy of force application; Will be evaluated by the simulated shot accuracy, horizontal displacement (X) and vertical displacement (Y).
6. Subjective parameters; in all time points, the volunteers will be asked to rate their level of pain sensation intensity (VAS sensory) and degree of unpleasantness (VAS affective) in the shoulders and other load bearing sites, as well as ratings of perceived exertion (RPE). All subjective parameters will be assessed using visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

Healthy medical status, fit (regular physical activity > 3 times weekly) men Previous experience with heavy backpack carriage Age: 18-35

Exclusion Criteria:

Heavy load carrying activity in the past 48 hr

Known diseases or medical conditions that may interfere with the study, of:

Musculoskeletal system Nervous system Cardiovascular system Vascular disease

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Neural performance of upper limb as measured by light touch sensitivity treshold | 1 hour
Neural performance of upper limb as measured by Thermal sensation treshold | 1 hour
Vascular performance of upper limb as measured by photoplethysmography of the index finger | 1 hour

SECONDARY OUTCOMES:
Motor function of upper limb as measured by force application of the index finger | 1 hour